CLINICAL TRIAL: NCT03166176
Title: SAMSUNG MEDICAL CENTER
Brief Title: Phase II Trial of Vistusertib（AZD2014） Single Agent in TSC1or 2 Null or TSC 1/2 Mutation Solid Cancer Patients Refractory to Standard Chemotherapy
Acronym: TSC1/2_SC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-05-096
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — vistusertib

STUDY DESIGN:
Intervention Model Description: Vistusertib(AZD2014) 50mg BD continuous schedule of a 28 day cycle
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Vistusertib(AZD2014) — vistusertib(AZD2014) is selective inhibitor of mTOR kinases and inhibits signalling of both mTOR complexes, mTORC1 and mTORC2.
  Other Names: AZD2014

SUMMARY:
Patients with TSC1/2 mutated refractory solid cancer will receive vistusertib(AZD2014) monotherapy. Study-arm is composed of 27 patients. Vistusertib(AZD2014) 50mg BD continuous schedule of a 28 day cycle as a monotherapy

DETAILED DESCRIPTION:
Patients with TSC1/2 mutated refractory solid cancer will receive vistusertib(AZD2014) monotherapy. Study-arm is composed of 27 patients.

Vistusertib(AZD2014) 50mg BD continuous schedule of a 28 day cycle as a monotherapy Tumour evaluation using RECIST 1.1 will be conducted at screening (within 28 days prior to first dose) and every 8 weeks relative to the date of first dose, up to week 40, then every 16 weeks until objective disease progression (within a window of +/- 7 days of the scheduled date).

Study treatment will be continued until objective disease progression (unless other criteria for treatment discontinuation are met). Patients may continue vistusertib(AZD2014) beyond progression (according to RECIST 1.1), at the discretion of the investigator if they are clinically benefiting from the treatment and they do not meet any other discontinuation criteria.

If a patient discontinues study treatment prior to disease progression, they should continue to be assessed using RECIST 1.1 until disease progression and then followed up for survival.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced solid cancers (including histologically or cytologically documented gastric cancer, colorectal cancer, hepatoma, biliary tract cancers, pancreatic cancer and rare cancers.) that has progressed after standard chemotherapy.
2. Provision of tumor sample (from either a resection or biopsy)
3. Patients with TSC1or 2 null or TSC 1/2 mutation through IHC.
4. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥9.0 g/dL (transfusion allowed)
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) > 3 x 109/L
   * Platelet count ≥100 x 109/L (transfusion allowed)
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
   * Serum creatinine ≤1.5 x institutional ULN

Exclusion Criteria:

1. Any previous treatment with PIK3CA, AKT or mTOR inhibitor or agents with mixed PI3K / mTOR activity.
2. For vistusertib(AZD2014):

   Exposure to potent or moderate inhibitors or inducers of CYP3A4/5 if taken within the stated washout periods before the first dose of study treatment With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.
3. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Objective reponse rate (ORR) by RECIST 1.1 | 12months
  To investigate the efficacy and safety of vistusertib(AZD2014) single agent as salvage therapy in patients with TSC1or 2 null or TSC 1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea